CLINICAL TRIAL: NCT01491399
Title: Study of Recombinant Human Bone Morphogenetic Protein-2 and Absorbable Collagen Sponge With the CORNERSTONE-SR™Allograft Ring and ATLANTIS™ Anterior Cervical Plate System in Treatment of Patients With Degenerative Cervical Disc Disease
Brief Title: INFUSE™ BONE GRAFT/CORNERSTONE-SR™ Allograft Ring/ATLANTIS™ Anterior Cervical Plate- Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-9702 Cornerstone ACDF pilot
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Cervical Disc Disease
MeSH Terms: interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- INFUSE™ Bone Graft/CORNERSTONE-SR™ (Experimental)
  Interventions: Device: INFUSE™ Bone Graft/CORNERSTONE-SR™ /ATLANTIS™
- Autogenous bone/CORNERSTONE-SR™ (Active Comparator)
  Interventions: Device: Autogenous bone/CORNERSTONE-SR™ /ATLANTIS™

INTERVENTIONS:
Device: INFUSE™ Bone Graft/CORNERSTONE-SR™ /ATLANTIS™ — Cornerstone-SR™ allograft bone containing recombinant human Bone Morphogenetic Protein (rhBMP-2) soaked into an absorbable collagen sponge (ACS) used in conjunction with ATLANTIS™ anterior cervical plate system.
  Other Names: recombinant human Bone Morphogenetic Protein-2; Infuse
  Arms: INFUSE™ Bone Graft/CORNERSTONE-SR™
Device: Autogenous bone/CORNERSTONE-SR™ /ATLANTIS™ — Cornerstone-SR™ allograft bone packed with autogenous iliac crest bone graft used in conjunction with ATLANTIS™ anterior cervical plate system.
  Other Names: Autograft
  Arms: Autogenous bone/CORNERSTONE-SR™

SUMMARY:
The purpose of this clinical trial is to assess the safety and effectiveness of the Investigational implant as compared to the Control implant in the treatment of patients with one level or two adjacent levels of cervical symptomatic degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical disc disease defined as: intractable radiculopathy and/or myelopathy with at least one of the following items producing symptomatic nerve root and/or spinal cord compression which is documented by diagnostic imaging procedures:

   * herniated disc;
   * osteophyte formation;
   * decreased disc height;
   * thickening of ligamentous tissue;
   * disc degeneration; and/or
   * facet joint degeneration.
2. Has preoperative Neck Disability Index score >= 30;
3. C2-C3 disc to C7-Tl disc level(s) of involvement.
4. One or two adjacent levels requiring fusion;
5. No previous surgical intervention at the involved fusion level(s);
6. Unresponsive to nonoperative treatment for approximately six weeks or has the presence of progressive symptoms or signs of nerve root or spinal cord compression in face of continued nonoperative management;
7. Age > 18 years at time of surgery;
8. Is female of child-bearing potential, who is not pregnant or nursing, and who agrees to not get pregnant for 1 year following surgery;
9. Willingness to comply with study plan and sign the consent form.

Exclusion Criteria:

1. Has cervical spinal condition requiring surgical treatment other than symptomatic cervical disc disease at the involved level(s).
2. Has been previously diagnosed with osteopenia, osteoporosis, or osteomalacia to a degree that anterior plating would be contraindicated.
3. Has presence of spinal metastases.
4. Has overt or active bacterial infection, either local or systemic.
5. Has fever (temperature > 101°F oral) at the time of surgery.
6. Has a documented titanium alloy allergy or intolerance.
7. Is mentally incompetent. If questionable, obtain psychiatric consult.
8. Is a prisoner.
9. Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug usage.
10. Has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of spinal fusion surgery (e.g., steroids or methotrexate), excluding routine perioperative anti-inflammatory drugs.
11. Has a history of autoimmune disease (Systemic Lupus Erythematosus or Dermatomyositis).
12. Has a history of exposure to injectable collagen implants.
13. Has a history of hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen.
14. Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following rhBMP-2/ACS implantation.
15. Has received any previous exposure to any/all BMP's of either human or animal extraction.
16. Has a history of allergy to bovine products or a history of anaphylaxis.
17. Has history of endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers- Danlos syndrome, or osteogenesis imperfecta).
18. Has a condition which requires postoperative medications that interfere with fusion, such as steroids, excluding routine perioperative anti-inflammatory drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 1999-09; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Fusion | 24 month
  Fusion is defined as:
  * No evidence of motion as defined by: less than 4° difference in angular motion between flexion and extension as seen on the lateral flexion/extension radiographs.
  * No radiolucency greater than 2mm of thickness covering more than 50% of superior or inferior graft surface.
  * Evidence of bridging trabecular bone.
Pain/Disability Status | 24 month
  The self-administered Neck Disability Index will be used. Success for each individual patient will be defined as pain/disability improvement postoperatively according to the following definition: Preoperative Score - Postoperative Score >= 15
Neurological Status | 24 month
  Neurological status will be assessed preoperatively and postoperatively using a comprehensive neurological status scale.

SECONDARY OUTCOMES:
Time to fusion | 24 month
Hip (Donor Site) Pain | 24 month
General Health Status (SF-36) | 24 month
Pain Status (neck pain, arm pain) | 24 month
Patient Satisfaction | 24 month
Patient Global Perceived Effect | 24 month